CLINICAL TRIAL: NCT07080879
Title: Clinical Study on the Advantages and Disadvantages of Linear Anastomat and Tubular Anastomat in Gastrointestinal Anastomosis During Radical Gastrectomy for Distal Gastric Cancer
Brief Title: The Advantages and Disadvantages of Linear Anastomat and Tubular Anastomat in Radical Gastrectomy of Distal Gastric Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STAPLER01
Record Dates: First submitted 2023-04-09; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-03

CONDITIONS: Gastric Cancer
Keywords: Linear Anastomat and Tubular Anastomat; Distal radical gastrectomy; Gastroenterostomy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Linear Anastomat Group (L Group) (Experimental): The duodenum and distal stomach were separated by linear anastomat at the planned tangents, and the specimens were taken out to confirm the safe cutting edge.The two arms of the linear anastomat were extended into the posterior wall of the duodenum and small openings at the stump of the greater curvature of the stomach respectively for cutting closure, and then the common openings were closed with the linear anastomat.
  Interventions: Device: Linear Anastomat
- Tubular Anastomat Group (C Group) (Active Comparator): The duodenum and distal stomach were separated by tubular anastomat at the planned tangents, and the specimens were taken out to confirm the safe cutting edge.The two arms of the tubular anastomat were extended into the posterior wall of the duodenum and small openings at the stump of the greater curvature of the stomach respectively for cutting closure, and then the common openings were closed with the tubular anastomat.
  Interventions: Device: Tubular Anastomat

INTERVENTIONS:
Device: Linear Anastomat — The product registration certificate numbers of linear anastomat is Su Wei registered 20202021581.
  Arms: Linear Anastomat Group (L Group)
Device: Tubular Anastomat — The product registration certificate numbers of tubular anastomat is Su Wei registered 20182020305.
  Arms: Tubular Anastomat Group (C Group)

SUMMARY:
The goal of this clinical trial is to observe and compare the short-term complications, long-term survival and quality of life of linear anastomat and tubular anastomat during digestive tract reconstruction after resection of distal gastric cancer.

Participants will receive a linear anastomat or tubular anastomat for digestive tract reconstruction during distal gastrectomy gastroenterostomy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≤ 18 years old ≤75 years old;
2. The primary gastric lesions were diagnosed as gastric adenocarcinoma (papillary adenocarcinoma pap, tubular adenocarcinoma tub, mucinous adenocarcinoma muc, sig-ring cell carcinoma, and poorly differentiated adenocarcinoma por) by gastroscopic biopsy.
3. The patient was clinically diagnosed with gastric cancer (in line with clinical signs of gastrointestinal reconstruction after distal subtotal gastrectomy for gastric cancer);
4. Implantation metastasis without peritoneum (confirmed by laparoscopic exploratory surgery);
5. It is estimated that R0 results can be obtained after D2 radical resection of distal gastric cancer (also applicable for multiple primary lower cancers);
6. Karnofsky score ≥60 points;
7. Preoperative ASA score: I, II, or III; 8。 Routine blood examination (no transfusion within the past 14 days) : HB≥90g/L;ANC ≥1.5×109/L;PLT ≥80×109/L；

9. Blood biochemical examination: BIL <1.5 times the upper limit of normal value (ULN);ALT and AST<2.5× ULN;Crea≤1 x ULN.

Exclusion Criteria:

1. Previous history of upper abdominal surgery (including gastric ESD/EMR, except laparoscopic cholecystectomy);
2. History of acute pancreatitis;
3. Preoperative imaging examination indicated fusion of enlarged lymph nodes (maximum diameter >3cm);
4. Gastric cancer patients who have received neoadjuvant therapy;
5. History of other malignant diseases within the past 5 years;
6. History of unstable angina pectoris, myocardial infarction, cerebral infarction, or cerebral hemorrhage within the past 6 months;
7. History of continuous systemic corticosteroid therapy in the past 1 month;
8. Concurrent surgical treatment for other diseases is required;
9. Patients with gastric cancer complications (bleeding, perforation) requiring emergency surgery;
10. Pyloric obstruction;
11. Lung function test FEV1< 50% of the expected value;
12. Pregnant or lactating women;
13. Suffers from severe mental illness;
14. Participate in other clinical studies at the same time;
15. Refused to sign the first round of study informed consent;
16. Unable or unwilling to comply with research requirements;
17. Patients with PD after neoadjuvant chemotherapy and unable to undergo distal gastrectomy;
18. Patients undergoing emergency surgery due to tumor bleeding, perforation and obstruction during chemotherapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Intraoperative Splenic Laceration | Perioperative period
  The number and percentage of participants experiencing splenic laceration during surgery.
Incidence of Positive Incisal Margin | Perioperative period
  The number and percentage of participants with a positive incisal margin after tumor resection.
Incidence of Anastomosis Failure | Perioperative period
  The number and percentage of participants experiencing anastomosis failure during surgery.

SECONDARY OUTCOMES:
Change in Procalcitonin Levels | Perioperative period
  The mean and standard deviation of procalcitonin (pg/mL or ng/mL) measured at designated time points (e.g., pre-operation, 1st post-operative day, 3rd post-operative day).
Change in C-Reactive Protein Levels | Perioperative period
  The mean and standard deviation of C-reactive protein (mg/L) measured at designated time points (e.g., pre-operation, 1st post-operative day, 3rd post-operative day).
Change in TNF-α Levels | Perioperative period
  The mean and standard deviation of TNF-α (pg/mL) measured at designated time points (e.g., pre-operation, 1st post-operative day, 3rd post-operative day).
Change in Interleukin-6 Levels | Perioperative period
  The mean and standard deviation of the percentage of CD3+, CD4+, CD8+, and NK cells among total lymphocytes, measured at designated time points (e.g., pre-operation, 1st post-operative day, 3rd post-operative day).
Health-Related Quality of Life assessed by EORTC QLQ-C30 Overall Score | 3 years
  The mean and standard deviation of the overall global health status/quality of life score from the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30), ranging from 0 to 100, with higher scores indicating better quality of life.
Disease-Specific Quality of Life assessed by EORTC QLQ-STO22 Score | 3 years
  The mean and standard deviation of relevant symptom scales and functional scales from the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Stomach Module (EORTC QLQ-STO22).

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital, Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided